CLINICAL TRIAL: NCT05484167
Title: Placebo-Controlled Cross-Over Pilot Trial of Natesto Testosterone Nasal Gel on Demand for Hypogonadal Men With Sexual Dysfunction Using Daily Phosphodiesterase-5 Inhibitor
Brief Title: Natesto Testosterone Nasal Gel for Hypogonadal Men
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: They study lost funding and decided to close the study down.
Sponsor: University of Utah (Other)
Collaborators: Acerus Pharmaceuticals Corporation (Industry)
Responsible Party: Principal Investigator, Jim Hotaling, Principal Investigator, University of Utah
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 00144770
Record Dates: First submitted 2022-06-09; First posted 2022-08-02 (Actual); Last update posted 2022-12-21 (Actual); Status verified 2022-12

CONDITIONS: Erectile Dysfunction; Sexual Dysfunction
MeSH Terms: conditions — Erectile Dysfunction; Sexual Dysfunction, Physiological

STUDY DESIGN:
Intervention Model Description: The patient crosses over at 90 days
Who Masked: Participant, Investigator
Masking Description: Double-Blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Natesto (Active Comparator): Natesto™ is a testosterone nasal gel that is FDA approved to treat low testosterone. It delivers testosterone through the nasal passages and it is then absorbed into the blood stream. The nasal pump is placed at the opening of each nostril and then the participant would press down on the nasal pump to apply the gel. Each application takes about 10 seconds and the nasal pump applies a thin layer of gel that absorbs through the lining of the nose.
  Interventions: Drug: Natesto Nasal Product
- Placebo (Placebo Comparator): This study involves a placebo. The placebo will look like the Natesto™ nasal pump and will contain a nasal gel, but without any active ingredients.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Natesto Nasal Product — Nasal Gel used for 90 days then crossed over to placebo gel
  Other Names: Natesto Nasal Gel
  Arms: Natesto
Drug: Placebo — A nasal gel with no active ingredients
  Arms: Placebo

SUMMARY:
To determine if testosterone deficient men who are using daily Tadalafil (a phosphodiesterase-5 Inhibitor), will have a significant improvement in erectile function and satisfaction with erectile dysfunction treatment when using on-demand Testosterone Nasal Gel (TNG) prior to sexual activity compared to placebo.

DETAILED DESCRIPTION:
The purpose of this study is to determine if testosterone deficient men whose primary symptom is erectile dysfunction, who are using daily Tadalafil (a phosphodiesterase-5 Inhibitor), will have a significant improvement in erectile function and satisfaction with erectile dysfunction treatment when using on-demand Testosterone Nasal Gel (TNG) prior to sexual activity compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and provide written informed consent for the study.
* Ability to read and complete electronic questionnaires in English.
* Adult males between the ages of 18-64 years
* Mild-moderate ED based on SHIM score between 8-21 at study entry
* Ability to take daily Tadalafil
* Ability to undergo venipuncture
* Ability to provide ejaculated semen sample
* Stable female sexual partner with sexual activity at least 1-3 times/month
* Hypogonadism defined as two (one done as SOC within the last 6 months and one done at the time of screening) early morning total testosterone lab values <300

Exclusion Criteria:

* Morbid Obesity - BMI >35
* History of Diabetes (HBA1c >6.0)
* Hematocrit < 35% or > 54% at study entry
* Concurrent or Prior use of other exogenous testosterone or hormone therapy (SERM, aromatase inhibitor, gonadotropins) within the last 3 months.
* Concurrent use of other prescription medications for ED including PDE5 inhibitors, intracavernosal injection therapy, urethral suppositories
* Concurrent use of nitrates in any form
* History of pelvic radiation
* Spinal cord injury
* Any progressive neurologic disease (Alzheimer's, Parkinson's, multiple sclerosis, etc).
* History of penile prosthesis
* History of prostatectomy
* History of transurethral resection of prostate
* History of stroke or myocardial infarction within the past 6 months
* History of congestive heart failure
* History of untreated obstructive sleep apnea
* History of liver disease (Serum transaminases > 2.5 times upper limit of normal)
* History of chronic kidney disease (GFR<60 or Serum Cr >2)
* History of, current or suspected, prostate (abnormal DRE or elevated PSA >4.0) or breast cancer.
* History of azoospermia or oligospermia (<15 million/ml)
* History of vasectomy
* History of Priapism
* History of Polycythemia Vera
* Receipt of any investigational product within 4 weeks of study enrollment
* Recurrent upper respiratory or sinus infection (>3 times/month for >6 months)
* Recurrent epistaxis (>3 times/month for >6 months)

Ages: 18 Years to 64 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — The study involves a diagnosis of Erectile Dysfunction. Therefore, all patients must have a penis, and this diagnosis.
Enrollment: 0 (Actual)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2024-01-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Comparison of Erectile Function and Sexual Intercourse Satisfaction Total Scores Recorded at Baseline and End of Study. | At Baseline and at the end of the study (Day 180)
  The primary endpoint of the study will be mean change in erectile function and satisfaction with sexual intercourse using the validated SHIM questionnaire. This questionnaire has been used extensively in clinical trials evaluating PDE5i for ED and is also used very commonly in the clinical practice. The SHIM Is a 5 item questionnaire that assesses the ability to get and maintain an erection sufficient for intercourse (Q1-Q4) and Q5 which assesses patient satisfaction. Each question is scored 0 to 5 with a total maximum score of 25.
  The investigators will look at the answers to all 5 questions and a higher score is interpreted as a better outcome.

SECONDARY OUTCOMES:
Comparison of Sexual Function Scores Recorded at Baseline and End of Study | At Baseline and at the end of the study (Day 180)
  Secondary outcomes will include a comparison of answers to question #2 in the Sexual Encounter Profile (SEP): Was the participant able to insert the penis into the partner's vagina? This is a question asked at baseline and at the end of the study. Answers are recorded as Yes or No and Yes is interpreted as a better outcome.
Comparison of Erection Success Recorded at Baseline and End of Study | At Baseline and at the end of the study (Day 180)
  Secondary outcomes will include a comparison of answers to question #3 in the Sexual Encounter Profile (SEP): Did the participant's erection last long enough to have successful intercourse? This is a question that will be asked at baseline and at the end of the study. Answers are recorded as Yes or No and Yes is interpreted as a better outcome.
Comparison of Treatment Satisfaction Total Scores at Baseline and End of Study | At Baseline and at the end of the study (Day 180)
  Secondary outcomes will include a comparison of the total score for the Treatment Satisfaction Questionnaire for Medication (TSQM-9) at baseline and again at the end of the study.
  The TSQM-9 scale is descriptive in nature and includes the following scales such as:
  1. Very satisfied
  2. Somewhat satisfied
  3. Neither satisfied nor dissatisfied
  4. Somewhat dissatisfied
  5. Very dissatisfied
  Higher scores are considered as a better outcome.
Comparison of Erectile Dysfunction Inventory of Treatment Satisfaction Total Scores at Baseline and End of Study | Baseline and at the end of the study (Day 180)
  Secondary outcomes will include a comparison of the total score for the Change in Erectile Dysfunction Inventory of Treatment Satisfaction (EDITS) at baseline and again at the end of the study. The EDITS scale is descriptive in nature and includes the following scales such as:
  1. Very satisfied
  2. Somewhat satisfied
  3. Neither satisfied nor dissatisfied
  4. Somewhat dissatisfied
  5. Very dissatisfied
  Higher scores are considered as a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: James Hotaling, MS, MS, Principal Investigator — University of Utah, Division of Urology, Department of Surgery
Locations (1):
- University of Utah, Division of Urology, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No